CLINICAL TRIAL: NCT04160845
Title: Compression of Non-invasive Forehead Skin Temperature to Core Temperature in Cardiac Surgery
Brief Title: Non-invasive Forehead Skin Temperature in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor Anesthesiology, Konkuk University Medical Center
Other Study IDs: 2019-11-008
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac surgery — cardiac surgery with hypothermic cardiopulmonary bypass

SUMMARY:
This study is to see if the zero-heat-flux (ZHF) thermometry monitoring in cardiac surgery with moderate hypothermic cardiopulmonary bypass differs from Temp-NP, which reflects central body temperature 30 minutes after the end of the cardiac surgery.

DETAILED DESCRIPTION:
This study is a single organ, prospective study of patients who are scheduled to perform cardiopulmonary surgery to compare noninvasive skin temperature attached to the forehead with core temperature after cardiopulmonary bypass in cardiac surgery.

anesthesia induction and maintenance use standard systemic anesthesia protocols using propofol-remifentanil-rocurium. Even before inducing anesthesia, it will start monitoring ECGs, noninvasive blood pigmentation, local cerebral oxygen saturation, blood pressure and heart rate.

After anesthesia induction and intraperitoneal intubation, the Temp-NP Hardness Ultrasound and Cardiac Output Monitoring through pulmonary artery catheter are initiated.

Before and after cardiopulmonary bypass, adjust the respiration rate of FiO2 04-0.5 so that the end tidal CO2 is 35-40 mmHg. Apply a positive end-expiratory pressure of 8 mmHg at the end of the period.

For surgery, heparin 3 mg/kg is administered, cardiopulmonary system is operated at medium-low body temperature, cardiopulmonary system is administered, and heart surgery is initiated from a cardiac standstill state. After the heart valve and coronary artery transplantation period, warm up to raise body temperature.

After recovering proper cardiac function, heparin is neutralized by administering 3 mg/kg of protamine and weaning from the cardiopulmonary bypass by administering inotropic agents.

After the anesthesia is finished, the patient is transferred to the intensive care unit in an intubated state, and is kept in isolation with dexmedetomidine until the tube is released.

The temperature monitoring of the sorcery starts the Temp-ZHF monitoring even before the anesthetic induction, and then the Temp-NP and Temp-PAC monitoring after the induction. Temp-NP monitoring devices are removed after surgery, but Temp-ZHF and Temp-PAC monitoring are also maintained in intensive care units after surgery.

The objectives of the study are as follows. primary goal Temp-ZHF vs. Temp-NP 30 minutes after cardiopulmonary bypass. secondary goal

1. After 30 minutes of anesthesia flow, there is a comparison between Temp-ZHF and Temp-NP.
2. It is compared to Temp-ZHF and Temp-PAC after 30 minutes of anesthesia.
3. Compared to Temp-ZHF and Temp-NP 30 minutes after cardiopulmonary bypass.
4. Compared to Temp-ZHF and Temp-PAC 30 minutes after cardiopulmonary bypass
5. 30 minutes after surgery, compared to Temp-ZHF and Temp-PAC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients over 19 years of age who are scheduled to undergo cardiac surgery are expected to apply cardiopulmonary bypass.
* 2. Patients Signed to Participate in Research

Exclusion Criteria:

* 1 Patient who refuses to sign consent form
* 2. Under 19 Criteria for exclusion during research

  1. In case a patient who decides to participate in a study refuses to make a decision or reverses (rejects) a decision after participation
  2. Patients who fail to perform Temp-NP surveillance during heart surgery
  3. Deep hypothermia patients
  4. Continuing the study is detrimental to the welfare of the study subjects

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 19 years of age who are scheduled to undergo cardiac surgery are expected to apply cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2020-09-02 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
comparison of skin temperature and nasopharyngeal temperature | 30 minutes after cardiopulmonary bypass
  comparison of Temp-ZHF vs. Temp-NP after cardiopulmonary bypass

SECONDARY OUTCOMES:
comparison between skin temperature and PA catheter temperature | 30 minutes after cardiopulmonary bypass
  comparison between Temp-ZHF and Temp-PAC 30 minutes after cardiopulmonary bypass

IPD SHARING:
Plan to Share IPD: No